CLINICAL TRIAL: NCT02452788
Title: Effectiveness of Pharmaceutical Care in Ambulatory Hemodialysis Patients: a Randomized Controlled Pilot Study
Brief Title: Pharmaceutical Care in Ambulatory Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Moinhos de Vento (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: AMhem-01
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Medication Adherence; Chronic Renal Diseases; Renal Failure Chronic Requiring Hemodialysis
MeSH Terms: conditions — Medication Adherence; Renal Insufficiency, Chronic | interventions — Pharmaceutical Services

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Intervention (Other): Pharmaceutical care with educational intervention provided by a pharmacist to ambulatory hemodialysis patients
  Interventions: Other: Pharmaceutical care
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Other: Pharmaceutical care — Pharmacist-provided education on medication adherence in hemodialysis patients.
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate the effectiveness of pharmaceutical care, compared to usual care, in improving medication adherence behaviour of ambulatory hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more
* Chronic renal patients undergoing regular hemodialysis
* Receiving their scheduled medications (at least one drug)

Exclusion Criteria:

* Unable to answer the questionnaire or to sign the informed consent form
* Inability to obtain prescription drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | one month
  High adherence according to the Brief Medication Questionnaire

SECONDARY OUTCOMES:
Quality of life | one month
  Quality of life will be evaluated with EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lisiane F Leal, MBA, Principal Investigator — Hospital Moinhos de Vento
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil